CLINICAL TRIAL: NCT07358091
Title: Investigation of Flexibility, Strength, and Posture in Women Practicingr Reformer Pilates Across Different Age Groups"
Brief Title: Investigation of Flexibility, Strength, and Posture in Women Practicing Reformer Pilates Across Different Age Groups"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-78097791-0204927
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer Pilates (Experimental): reformer pilates- 46-60 age
  Interventions: Other: Reformer Pilates
- reformer pilates (Experimental): reformer pilates- 18-45 age
  Interventions: Other: Reformer Pilates

INTERVENTIONS:
Other: Reformer Pilates — Reformer Pilates is a low-impact exercise method performed using spring-based equipment that aims to improve muscle strength, flexibility, core stability, and postural control in women aged 18-46 through controlled and precise movements.
Other: reformer pilates — Reformer Pilates is a low-impact exercise method performed using spring-based equipment that aims to improve muscle strength, flexibility, core stability, and postural control in women aged 46-65 through controlled and precise movements.

SUMMARY:
"Investigation of Flexibility, Strength, and Posture in Women Practicing Regular Reformer Pilates Across Different Age Groups"

DETAILED DESCRIPTION:
"Investigation of Flexibility, Strength, and Posture in Women Practicing Regular Reformer Pilates Across Different Age Groups"

ELIGIBILITY:
Inclusion Criteria

* Female participants aged 18-65 years
* Regular participation in Reformer Pilates exercises
* Voluntary participation with signed informed consent
* No medical condition preventing participation in the assessment and testing procedures

Exclusion Criteria

* Pregnancy
* History of spinal surgery within the last 6 months
* Presence of neurological conditions affecting mobility (e.g., Parkinson's disease)
* Presence of chronic systemic diseases (e.g., cancer, diabetes)
* Severe pain-related movement limitation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 38 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Flexibility Assessment | 5 weeks
  Flexibility was assessed using the Sit-and-Reach Test
Sørensen Test | 5 weeks
  This test is a widely used and reliable method for assessing the isometric endurance of the erector spinae muscles
Trunk Flexor Endurance Test | 5 weeks
  Participants were positioned in a seated posture with the trunk inclined at 60°, the knees flexed at 90°, and the arms placed either across the chest or behind the head. Participants were instructed to maintain their trunk at this angle for as long as possible, and the endurance time was recorded in seconds using a stopwatch. This test was conducted to assess the isometric endurance of the trunk flexor muscles, particularly the rectus abdominis and iliopsoas muscles
Lateral Bridge (Side Bridge) Test | 5 weeks
  Participants were positioned in a side-lying posture, supporting their body on the lower arm and the lateral aspect of the feet, maintaining the trunk in a straight line. The upper arm was placed on the hip, and participants were instructed to hold this position for as long as possible. The endurance time was recorded in seconds using a stopwatch. This test is a commonly used method to assess the isometric endurance of the oblique muscle groups and the quadratus lumborum muscles
Muscle Strength and Body Composition Assessments | 5 weeks
  In this study, the Visbody 3D body analysis system was used to evaluate participants' body composition and postural characteristics through millimetric three-dimensional scanning. The system provided segmental muscle mass analysis for the upper extremities, lower extremities, and trunk, enabling a detailed assessment of the relationship between muscle distribution and strength and endurance outcomes. In addition to body composition parameters such as body fat, fat-free mass, BMI, and visceral fat, postural variables including spinal alignment, shoulder and pelvic symmetry, pelvic tilt, and shoulder joint angles (abduction and flexion) were assessed. Overall, Visbody supplied comprehensive, multidimensional data that supported functional test results and enhanced measurement reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No